## **Official Title:**

Posterior slab vs total contact cast in diabetic foot ulcers: a randomised controlled trial

NCT number: Not received yet

**Document date: 31/07/2025** 

### PROTOCOL ILSS/EC/0012-DFU/2022

# POSTERIOR SLAB VS TOTAL CONTACT CAST IN DIABETIC FOOT ULCERS: A RANDOMISED CONTROLLED TRIAL

ILS Hospital, DD-6, Sector-1, Salt Lake, Kolkata-700064, West Bengal

### **Table of Contents**

| 1. | Affiliation | Page 2 |
|-----|--------------------------------|---------|
| 2. | Introduction | Page 3 |
| 3. | Aim and Objectives | Page 3 |
| 4. | Inclusion & Exclusion criteria | Page 3 |
| 5. | Materials and Methods | Page 4 |
| 6. | Outline of time plans | Page 4 |
| 7. | Statistical analysis | Page 4 |
| 8. | Ethics | Page 4 |
| 9. | Sources of funding | Page 4 |
| 10. | Primary References | Page 5 |
| 11. | <b>Copy of Consent Forms</b> | Page 6 |
| 12. | Copy of Foot History File | Page 9 |
| 13. | CV, MRC & GCP | Page 17 |

### 1. AFFILIATIONS

### **Research Institute**

ILS Hospital, Salt Lake.

Address: DD-6, Sector 1, Salt Lake City, Kolkata-700064

Principal Investigator-cum-Guide : Dr. Ghanshyam Goyal

Address: ILS Hospital, Salt Lake,

DD-6, Sector 1, Salt Lake City, Kolkata-700064

Phone Number: +91-9830400450 Email: drgsgoyal@hotmail.com

**Co-Guide** : Dr. Rekha Srivastav

Address: ILS Hospital, Salt Lake,

DD-6, Sector 1, Salt Lake City, Kolkata-700064

Phone Number: +91-9831058704 Email: ins.rekha@gmail.com

#### 2. INTRODUCTION

There are three basic principles in the management of diabetic foot ulcer (DFU) – adequate debridement and infection control, adequate vascularity, and adequate offloading. Off-loading of the ulcer area is extremely important for the healing of neuropathic plantar ulcers. Total Contact Cast (TCC) remains the gold standard treatment of Diabetic Foot Ulcer (DFU). However, there are many practical problems associated with TCC, including local skin irritation, worsening of deformed toe nails, fungal infections, claustrophobia, joint rigidity, atrophy of the smaller foot muscles, postural instability and painful leg and calf muscles. So, TCCs are underutilized in clinical practice as they are technically difficult and time consuming to apply, relatively expensive and have low patient tolerance. Their use is also contraindicated in patients with infected or ischaemic ulcers. Posterior slab cast (PSC) is also a good offloading modality in neuropathic DFU. It can be more convenient and economical as a single slab can be used till complete healing is achieved. Thus may provide a lesser invasive way of immobilization of the foot in DFU.

#### 3. AIM & OBJECTIVES

Aim of this trial is to compare the efficacy of Posterior slab cast (PSC) with Total Contact cast (TCC) in terms of wound healing and foot related outcomes in patients having neuropathic planter diabetic foot ulcers in a tertiary care diabetic foot clinic.

#### 4. INCLUSION AND EXCLUSION CRITERIA

#### Inclusion criteria

- 1. Type 2 Diabetes Mellitus
- 2. Having solitary neuropathic plantar ulcer
- 3. Ulcer belonging to Wagner's grade 2 or 3

#### Exclusion criteria

- 1. Persons with bilateral DFUs
- 2. Peripheral vascular disease (ABI < 0.9)
- 3. Gout
- 4. steroid intake in the last three months,
- 5. Stage 4 & 5 chronic kidney disease with estimated glomerular filtration rate (eGFR) <30 ml/min/m2,
- 6. Bilateral foot involvement,

### 5. MATERIAL & METHODS

It is an open label randomized control trial. It will be done in ILS Hospital, Kolkata for a trial period of around 3 years.

Diabetic patients attending the foot clinic with plantar ulcer irrespective of age, sex, glycemic control, duration of diabetes, duration of ulcer and presence of infection will be considered for the study. At first patients will be randomly allocated to any one of two off-loading procedures using the randomization table: TCC or PSC. Those who will refuse TCC, will be shifted to PSC group. All patients will be followed up at the foot clinic once in two weeks' basis for device inspection, wound care and wound debridement as and when indicated. After the completion of treatment, all the patients will be followed up to 15 months from the initiation of treatment to identify any recurrence of ulcer.

Two outcome measures will be used. The primary outcome measure is healing of the ulcer after 8 months. The secondary outcome measure is to document which of the device is associated with comparatively better healing at 6 months.

### **6. OUTLINE OF TIME PLANS:**

Proposed date of starting research activity: January 2023

Expected duration of research activity: 1.5 years

Undertaking to provide interim report of the work halfway through it: Yes

Undertaking to provide full report of the work on completion: Yes

#### 7. STATISTICAL ANALYSIS:

Comparison will be done between the two groups. Continuous variables will be compared by t-tests and categorical variables by chi-square test. Baseline comparison will be made using chi-square tests and two-sample t-tests. Continuous variables will be expressed as mean (standard deviation). The differences in pertinent characteristics will be established with the use of t-test for independent samples. A two-sided p value of 0.05 was considered statistically significant.

### 8. ETHICS

01) Subject information brochure: Yes

02) Informed consent form: Yes

03) Statement of conflict of interest, if any: None

Publication-plans for the outcome (positive or negative) while maintaining the privacy and confidentiality of the study participants:

The privacy and confidentiality of the study participants will be maintained in all publications/reports originating from this study.

### 9. SOURCE(S) OF FUNDING:

Not Applicable

### 10. PRIMARY REFERENCES:

- 1) A mouldable fibreglass backslab device as a novel approach to offload chronic plantar foot ulcers: A retrospective observational audit; First published: 21 August, 2024,https://doi.org/10.1002/jfa2.70001
- 2) Li B, Lin A, Huang J, Xie J, Liu Q, Yang C, Zhang Z. Total contact casts versus removable offloading interventions for the treatment of diabetic foot ulcers: a systematic review and meta-analysis. Front Endocrinol (Lausanne). 2023 Sep 26;14:1234761. doi: 10.3389/fendo.2023.1234761. PMID: 37822605; PMCID: PMC10562689
- 3) A Comparative Study Between Total Contact Cast and Pressure-Relieving Ankle Foot Orthosis in Diabetic Neuropathic Foot Ulcers; Partha Pratim Chakraborty et al; Journal of Diabetes Science and Technology 2015, Vol. 9(2) 302 –308 © 2014 Diabetes Technology Society Reprints and permissions: sagepub.com/journalsPermissions.nav DOI: 10.1177/1932296814560788

#### 11. COPY OF THE CONSENT FORMS:

# POSTERIOR SLAB VS TOTAL CONTACT CAST IN DIABETIC FOOT ULCERS: A RANDOMISED CONTROLLED TRIAL

Study to be conducted by: Dept of Diabetology & Diabetic Foot Clinic, ILS Hospitals, Saltlake

You are being invited to participate in a clinical research trial. The following information is for you to understand why the research is being done and what it will involve. Please take time to read it carefully and discuss with friends, relatives and your family doctor if you wish. Please feel free to ask us if there is anything that is not clear or if you would like more information. Take time to decide whether or not you wish to take part. Please sign the Informed Consent Form only if you are fully satisfied with the information given to you and you understand the procedures involved in the study.

### What is the purpose of the trial?

Aim of this trial is to compare the efficacy of Posterior slab cast (PSC) with Total Contact cast (TCC) in terms of wound healing and foot related outcomes in patients having neuropathic planter diabetic foot ulcers in a tertiary care diabetic foot clinic.

### Why have I been chosen?

Diabetic patients having solitary neuropathic plantar ulcer have been chosen for the study. You have been selected because you have an foot ulcer and also satisfy the other selection criteria for the study.

### Do I necessarily have to take part?

No, it is up to you to decide whether or not to take part. If you decide to take part, you will be asked to sign a consent form. Even after you have decided to take part, you are still free to withdraw anytime you choose without giving us a reason. A decision to withdraw, or a decision not to take part, will not affect the quality of care you receive.

### What happens during the study?

If you agree to participate, no extra intervention will be done and neither any special drugs will be used. We will use the post-trial data generated for a clinical research purpose.

### Are there any other possible disadvantages of taking part?

No disadvantages since the data generated post-trial will be used for research purpose.

### Will my taking part in this study be kept confidential?

Yes. All data obtained from the study will be kept confidential. The data would be archived for an appropriate period. This data will be used only by authorized persons for scientific purposes.

### What will happen to the results of the study?

A study report will be finalized soon after the trial closes. This will be submitted to the ethics committee of the institute carrying out the study, and also to government authorities if needed. The results may be published in a scientific journal or discussed at a scientific forum. You will however, not be identified in any report / publication.

#### **Contact for further information:**

The doctors conducting this study can discuss it in more detail with you and reply to any query, when it arises. The contact persons are:

| Dr. Ghanshyam Goyal | Dr. Rekha Srivastav |
|--------------------------------------|---------------------------------|
| Principal Investigator | Co-Guide |
| ILS Hospital, Saltlake | ILS Hospital, Saltlake |
| DD-6, Sector-1, Salt Lake City, | DD-6, Sector-1, Salt Lake City, |
| Kolkata - 700064 | Kolkata - 700064 |
| Ph No:+91-983040450 | Ph No: +91-9831058704 |
| Email: drgsgoyal@hotmail.com | Email: ins.rekha@gmail.com |
| Principal Investigator - cum - Guide | Co-Guide |

Thank you for going through the Patient Information Sheet.

Should you decide to participate in this clinical study, we thank you for that too.

### INFORMED CONSENT FORM

# POSTERIOR SLAB VS TOTAL CONTACT CAST IN DIABETIC FOOT ULCERS: A RANDOMIED CONTROLLED TRIAL

| Patient's: Name: | Initials | Age | Sex | | _ |
|---|---|---|---|---|---|
| 1. I confirm that I have read and understood the informati-<br>the above study and have had the opportunity to ask quest | | | | [ | ] |
| 2. I understand that my participation in the study is volunt free to withdraw at any time, without having to give a reas without my medical care or legal rights being affected. | - | am | | ] | ] |
| 3. I understand that my data would be kept confidential be authorized by the Principal Investigator, the ethics commi where the study will be conducted and government drug rewill have access to my health records both in respect of the and further research that may be conducted in relation to it I agree to this access. However, I understand that my identifications are the study of | ttee of the inst<br>egulatory auth<br>e current stud<br>t. Even if I wit | ority<br>y<br>hdraw, | | | |
| revealed and confidentiality of information will be mainta | ined. | | | [ | ] |
| 4. I agree not to restrict the authorized use of any data or r From this study. | esuits that aris | se | | [ | ] |
| 5. I agree to voluntarily take part in the above study. | | | | [ | ] |
| Signature / Thumb impression of the subject: | | | | | |
| Date:Place: | | | | | |
| Study doctor's name: | | | | _ | |
| Study doctor's signature:Date: | Pla | ce: | | | |
| Mandatory where subject has provided thumb impress | sion: | | | | |
| Signature of the witness: | | | | | |
| Date:Place: | | | | | |
| Name & Address of the witness: | | | | | _ |
| Relation to the subject, if any: | | | | | _ |

### 12. COPY OF HISTORY FILE

# POSTERIOR SLAB VS TOTAL CONTACT CAST IN DIABETIC FOOT ULCERS: A RANDOMIED CONTROLLED TRIAL

# CASE REPORT FORMS TO BE FILLED AT THE TIME OF FIRST OP VISIT

| HOS | PITALS | | | res & o | | CLINIC<br>RM) | | | |
|---|---|---|---|---|---|---|---|---|---|
| Date | | | | | | | UHID I | No | |
| 1. Patien | t Details : | | | | | | | | |
| Name : | | | | | | Age : | | Sex : Ma | le / Fem |
| Address | : | | | | | | | | |
| Marital S | tatus : | | Rel | igion : | | Occu | pation : | | |
| Phone N | os. : | | | | Mo | bile No. : | | | |
| Refd. By | Dr. : | | | | Under | Consultant | Dr | | |
| | ic History : | | | | | ¢. | ** | 9 | |
| Age of O | nset : | | | Mode | of Onset : | Accidental | / Others | | |
| | | | | | | | 4 | | |
| Duration | Of diabetes | : | | Tre | atment Tak | en for DM∵: . | | | |
| Duration | Of diabetes | : | | Tre | atment Tak | en for DM∵: . | | | |
| Duration 3. Family | Of diabetes History of D | :<br>Diabetes. | | Tre | atment Tak | en for DM: | | | |
| Duration 3. Family | Of diabetes | i<br>Diabetes.<br>amily is suff | | Tre | atment Tak | en for DM: | | | |
| Duration 3. Family Is anyb | Of diabetes History of Dody in the fa | i<br>Diabetes.<br>amily is suff | fering from | Tre | atment Tak | en for DM: | | | |
| Duration 3. Family Is anyb | Of diabetes History of Dody in the fa | i<br>Diabetes.<br>amily is suff | fering from | Tre | atment Tak | en for DM: | | | |

Others ILS/OPD/AAC/2019/21

Heart Disease
Kideny Disease
Liver Disease
Asthma / COPD
Hypertensions
Chronic Infections



HbA1c

Others

## **DIABETES & OBESTTY CLINIC**



| Reason | Treatment (Surgical / Conse | ervative) | Dates |
|---|---|---|---|
| 5. Present History of | Diabetics : | | |
| A. Present Sympto | ms : | | |
| B. Treatment Recei | ivina now : | | |
| | 4 | | |
| | * | | |
| OHA + INSULI | N: | | |
| INSULIN: | | · | |
| ALTERNATIVE | MEDICINE : | | |
| ☐ NO MEDICINE | * | | |
| C. Any Symptoms ( | | | |
| f YES | ☐ HOSPITALISATION | DOMESTIC TRE | ATMENT |
| □ NO | | | |
| D. Recent B. Sugar | Values | | |
| Blood Sugar | Values | Date | |
| RBS | 8 | | |
| FBS | | | |
| PPBS | | e | |





E. Complication of Diabetes :

| | Present / Absent | Duration | Treatment received if any |
|--------|------------------|----------|---------------------------|
| Eye | | | |
| Kideny | | | |
| Heart | | | |
| Foot | | | |
| Nerves | | | |
| Others | | | |

| 6. For Female Patient : | | | | |
|---|---|---|---|---|
| Gravida | | Parity | H/O GDM | |
| Gynecological Problems (I | f Any) | | | |
| 7. Physical Examination : | • | | | |
| | | 1 | | |
| 1. Height: | Weight: | , BMI: | EBW: | |
| 2. Pulses : Rate : | | beats per min, Rhy | rthm : Regular / Irregular | |
| Radial | | | | |
| Brachial | | | , | |
| <ul><li>Carotid</li></ul> | • | | ¥ ** | |
| <ul><li>Femoral</li></ul> | 3 | | | |
| <ul><li>Dorsalis Pedis</li></ul> | <b>3</b> | | | ¥ |
| 3. Blood Pressure : Standing | ng : | mm of Hg; Supir | ne | mm of Hg |
| 4. Thyroid: | | 5. Oedema : | * | |
| 6. Respiratory System : | | 7. Cardio Va | scular System : | |
| 8. Abdomen : | | 9. Skin / Eye | <b>5</b> : | |
| 10. Central Nervous Syster | m: | 11. Others : | 4 e | |





| 8.Investigatio | n : | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | B-4 | | | | | |
| Туре | Dates | | | | | | | | | | |
| | | | <u> </u> | | | | | | | L | |
| BLOOD SUGAR | | | | | , | 1 | | <del></del> | | Γ | |
| FBS | | | | | | | | | - | | |
| PPBS | | | | | | | | | | | |
| RBS | | | | | | | | | | | - |
| Hb1Ac | L | L | | | <u> </u> | | L | L | <u> </u> | L | |
| RENAL | | | | | | т | 1 | | I | | |
| Urea | | | | , | | | | | | | |
| Creat. | | | | | | | | | | | |
| Micro albumin | | | | | | ` . | | <u>.</u> | | | |
| 24 Hr. Urine | | | | <u></u> | | | - | | | | |
| Protein | | | | | | - A.M | | | | | |
| Creatinine | | | | ļ | | | | | | | |
| Clearance | | | <u> </u> | | <u> </u> | EAT. | | | L., | | |
| BLOOD LIPIDS | | | 1 | | | | | | т | | T - |
| Cholestrol | | | | * | | | | | | | |
| Triglyceride | | | | | | · | | | | | |
| HDL | | | | | | | | | | | |
| LDL | | | | | | | | | | | |
| VLDL | | | | | | | | L | | <u></u> | <u> </u> |
| LFT | | | 4 | | _ | | | | | | |
| Bill (T) | to to | | (1) | | | | | | | | |
| Bill (D) | | | | | | | | | | | |
| Bill (I) | | | | | | | | | | | |
| Protien | | | | | | | | | | , | |
| Alb | * | | | | | 1 | | | | | |
| Glob . | | | | , | | | | | | | |
| SGOT | | | | | | 100 | | | | | |
| SGPT | | 3 | | | | | | | | | |
| Alk Ph. | | | | 8 6 | | | 70 - S | | | | |
| GGT | | | | | | | | | | | |
| Uric Acid | .: | 1. | | | | | | | : | | |
| HAEMOGRAM | · | | | | | | | | | | |
| Hb% | | ' | | | | - | | | | | |
| WBC | | | | | | | | | e , | | |
| DC | | | | | | | | i i | | | |
| ESR | | | | | | | | | | | |
| Plat. | | | | | | | | | | | |
| PCV | - | | 1 | | | | | | | 1/40 | |





| | | | | | | - | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Dates | | | | | | | | | | | |
| Albumin | | | | | | | | | | | |
| Glucose | | | | | | | | | | | |
| Ketone | | | | | | | 0 | | | | 8 |
| RBC | | | | | , | | | | | | |
| Leukocytes | | | | | | | | | | | |
| | | 1 | l— . | <u> </u> | • | | | | | 141 | |
| Т3 | | | 100 | | | | | | | | |
| T4 | | | | | | | | | | | |
| TS | | | | | | | | | | | |
| Calcium | | | | | | | | | 2.8 | | |
| | | <u> </u> | <del>L</del> | L | d | 3 | | | 2<br>1 | | |
| | | T | | | | | | | , | | |
| | | | | | | | | 1 | | 1. | |
| | | | | | | | | • . | | | ř |
| | · · | | | | | | | , | | | |
| | | | 1 | | | | | | | | |
| | | - 1 | | | | | | | | | |
| | | | - | | | | | | • | | . 6 |
| TYPES | | <del></del> | | | DATES | | | | | | <del></del> |
| | | Γ | <u> </u> | | | **** | | | | Γ | |
| RETINA | | 2 | | | | | | | | | |
| | | | | | 170 | | | | | | |
| X- RAY | <del>- </del> | | | | <b></b> | | | | | | |
| ECG | | | | - | | | | | | | |
| USG | <del>-</del> | | | | | | | | | | |
| ECHO | | | | | | | · · | | | | |
| Foot Examination | n : | | L | | | | | | | | |
| Monofilament : | <b></b> | | | | | | | | | | |
| Right : | | | | | | | | | - | | |
| Left : | | I. | <del></del> | <u> </u> | | | | | | | |
| VPT: | | | | | | | | | | | |
| Right: | | | | | | | | | | | |
| Hot & Cold Perc | Left : Hot & Cold Perception : | | | | | | | | | | |
| Right : | | | | | | | | | | <del></del> | |
| Left: | | | | | | | | | | | |
| ABI / DOPPLER | | 100 | 307 | | | | | | - | | |
| Right: | | | | | | | | | | | |





| DATE | FOLLOW UP COMPLAINTS | TREATMENT ADVICE |
|------|----------------------|-----------------------------------------|
| | | * · |
| | • | ,<br>~, |
| | l | |

| NAME: | AGE: | SEX: |
|----------------|------------------------------|------|
| ADDRESS: | | |
| MOB.NO: | REFFERING DR.: | |
| <u>MEDICAL</u> | <b>DIABETIC FOOT HISTORY</b> | |
| <u>HISTORY</u> | | 000 |
| | рт гт | |

| <u>MEDICAL</u> | <b>DIABETIC FOOT</b> | <b>DIABETIC FOOT HISTORY</b> | |
|---|---|---|---|
| HISTORY | | | |
| | | RT | LT |
| Duration of | Duration of Ulcer | | |
| Diabetes | | | |
| Duration of | Past H/O Ulcer | | |
| Hypertention | | | |
| Hight | H/O Amputation | | |
| Weight | Joint pain | | |
| BMI | Stiffness | | |
| Dyslipidemia | Dry skin | | |
| SMOKER | Numbness | | |
| CVD | Tingling/Pricking | | |
| CKD | Paresthesia | | |
| Blood Sugar | Claudication | | |
| HbA1C | Cramping | | |
| | Oedema | | |



# EXAMINATION OF FOOT INSPECTION

| | _ | | | | |
|----------|-----|----|--------------|-----|----|
| DRY SKIN | YES | NO | ABNORMAL | YES | NO |
| | | | SHAPE | | |
| FISSURE | YES | NO | NAIL LESION | YES | NO |
| DEFORMIT | YES | NO | LOSS OF HAIR | YES | NO |
| Y | | | | | |
| CALLUS | YES | NO | | | |

| <b>PALPATION</b> | НОТ | CO | LD | NORMA | 1 | 1 | | 1 1 |
|---|---|---|---|---|---|---|---|---|
| | | | | L | 1 | 1 | | 1 |
| RIGHT | | | | | Y = | 1 | | YEY |
| LEFT | | | | | | | | 1 . / |
| <b>FOOT PULSES</b> | RT | | | LT | 2 | 1 | , | 2 |
| DORSALIS | | | | | 5 | 3 | | (e) 1 Lb) |
| PEDIS | | | | | 6 | <b>3</b> 4 | 4 | |
| POTERIOR | | | | | | | | |
| TIBIALIS | | | | | | | | |
| <b>ASSESSMENT</b> | OF | | | RIGHT | RIGHT | LEFT | | LEFT |
| <b>NEUROPATHY</b> | <u>Y</u> | | | | | | | |
| MONOFILAME | NT | | | | | | | |
| VPT | | · | | | | | | |
| HCP | | | | • | | | | |

| VASCULAR | RIGHT | LEFT |
|--------------------|-------|------|
| <u>ASSESSMENT</u> | | |
| DORSALIS PEDIS | | |
| POSTERIOR TIBIALIS | | |
| BRACHIALIS | | |
| ABI | | |





## RADIOLOGICAL INVESTIGATION (X RAY FOOT)

RT:-LT:-

## **DESCRIPTION OF ULCER**

Location :-Size:-Base:-Margins:-

| Depth:- | | | | | | |
|--------------------|-----|----|----|------------------------|-------|---|
| CLINICAL DIAGNOSIS | | | | WEGNERS CLASSIFICATION | | |
| | YES | NO | | Grade-0 | | |
| NEUROPATH | | | | 1-Superficial | Ulcer | |
| Y | | | | _ | | |
| CHARCOT | | | | 2-Deep Ulcer | r | |
| FOOT | | | | _ | | |
| PVD | | | | 3-Osteomyelitis | | |
| INFECTED | | | | 4-Localized Gangrene | | |
| OTHERS | | | | 5-Extensive Gangrene | | |
| | • | | .~ | 270 | _ | • |

| OTTILLIA | | | | 5 Littonsi i C |
|--------------------|----------|-------|---|----------------|
| TREATMENT | | YE | S | NO |
| Callus and Corn Re | emoved | | | |
| Nail paring | | | | |
| I+D done | | | | |
| Pus for CS | | | | |
| Probing | | | | |
| Extensive debriden | nent | | | |
| Surgical Referral | | | | |
| Others | | | | |
| OFFLOADING T | ECHNIQUE | YE YE | S | NO |
| S K OFFLOADING | G | | | |
| OFFLOADING SH | ЮЕ | | | |
| TOTAL CONTAC | CT CAST | | | |
| INSTANT TCC | | | | |
| CUSTOM FOOTV | VEAR | | | |
| OTHERS | | | | |

### FOLLOW UP

## Specialised Medical Personnel Curriculum Vitae

| DR. GHANASHYAM GOYAL |
|---|
| SENIOR CONSULTANT - DIABETOLOGIST |
| PRINCIPAL INVESTIGATOR |
| ILS Hospltd DD·6, SEC-1 ,SALTLAKE,KOL-64 |
| MBBS-1984, MD-1988 |
| Director & Consultant Diabetologist & Diabetic Foot<br>Specialist, S.K. Diabetes Research and Education<br>Centre, Kolkata - February 2006 - till date |
| Consultant, Dept. of Internal Medicine and Head, Dept. of Dlabetology, ILS Hospital, Kolkata - January 2002 - till date |
| Consultant Physician & Diabetologist - Unit Head,<br>MRS Hospitals - January 1996 - 2002 |
| Consultant Physician & Diabetologist - MRS<br>Hospitals, Kolkata June 1991 - December 1995 |
| Chief Resident - Dept. of Internal Medicine - MRS<br>Hospitals, Kolkata - October 1988 - May 1991 |
| Quintiles Online GCP - 2011 |

| Relevant ClinIcal Trial and Research Experience | PRINCIPAL INVESTIGATOR: |
|---|---|
| including GCP Training: | A trial comparing the efficacy and safety of |
| mercang oci Trannig. | insulin degludec I liraglutide and insulin |
| | degludec in subject with type 2 diabetes. |
| | PRINCIPAL INVESTIGATOR: |
| | Efficacy and Safety of H0/03/03 10 ug in the |
| | treatment of Neuropathic Diabetic Foot |
| | Ulcers - A PHASE II TRIAL (a double |
| | · · |
| | blind placebo controlled ,Multicentre study) |
| | PRINCIPAL INVESTIGATOR: |
| | BIOCHAPERONE PDGF - BB - A |
| | phase I/II, multicentre, |
| | randomized,controlled, open label trial |
| | comparing the |
| | efficacy and safety of two dose regimens of |
| | BioChaperone POGF - BB to becaplermin |
| | gel for the treatment of diabetic foot ulcer. |
| | DIABESITY: Role of Insulin Detemir, an open label, |
| | observational, multicentric, randomized study in April |
| | 2008. |
| Other Activities Pertinent to Professional | <b>INSUTREAT:</b> A registry to study the effect |
| Qualifications | of changes of existing Insulin treatment in |
| | Inadequately controlled Type 2 diabetes patients |
| | till February 2007. |
| | The <b>IMPROVE:</b> study A multicentre, open |
| | label, non randomized, non interventional, |
| | observational, safety & effectiveness study in |
| | subjects using Biphasic Insulin Aspart 30 for |
| | t he treatment of DM in 2007. |
| Certifications and Licensures: | Diabetology research course in |
| (Optional) | genetics (Star Steno diabetes educatiori |
| | project} at Bangalore inAugJst, 2005. |
| | Advanced Dishetes & Endocrinology |
| | Advanced Diabetes & Endocrinology Precentorship at John Hopkin's University |
| | Preceptorship at John Hopkin's University, |
| | School of Medicine, Baltimore, USA in |
| | March 2008. |

Faculty & Trainer Staged Diabetes Management for Physicians, conducted by International Diabetes Centre.

Started the first Diabetic Foot Clinic of Kolkata & Eastern India in 2003

Regional Coordinator: "National Wound Care Project"(WOF DFSI)

Regiona Faculty - Certificate Course in Evidence Based Diabetes Management conducted by Public Health Foundation of India (PHFI)

Conducting Workshops on Diabetic Foot all across the country to inc ease awareness amongst Paramedics, Physicians and D1abetologists

Signature of Trial Site Staff/
Specialised Medical Personnel: 

| Ship | Date: 07 | Feb | 2022 | Yyyy | Yyyy | Signature of Trial Site Staff/ | Specialised Medical Personnel: | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship | Ship |

### NAME: DR REKHA BASAK SRIVASTAVA

E-MAIL ID: ins.rekha2@gma il.com

EDUCATIONAL QUALIFICATION: B Sc, BAMS

Clinical podiatrists and Chief Clinical Research Co ordinator - ILS Hospital, Kolkata

#### PROFESSIONAL TEAC HING EXPERIENCE TILL DATE:

- 1. Best paper presentation award in DFSI KOLKATA'2008
- 2. Master trainer of IDF Certified course- project HOPE (Indian diabetic educator project)
- 3. Chief of clinical podiatry program me, conducted workshops at different medical colleges under DFSI wound care project
- 4. Conducted workshops at different states under Diabetic Foot Education Programme (DFEP).
- 5. Conducting patient education programme for Diabetes and Diabetic foot every month at ILS HOSPITAL ,SALT LAKE.

### Working as Clinical Research Co ordinator:

- 1. A Phase III, Multicentre, Randomized, Parallel Group, Double Blinded and Control Group Clinical Trial to Assess the Effectiveness of Biochaperone PDGF-BB in the Treatment of Chronic Diabetic Foot Ulcer
- 2. A trial comparing the efficacy and safety of insulin degludec I liraglutide and insulin degludec in subject with type 2 diabetes.
- 3. Efficacy and Safety of H0/03/03 10 ug in the treatment of Neuropathic Diabetic Foot Ulcers A PHASE II TRIAL ( a double blind placebo controlled ,Multicentre study)
- 4. BIOCHAPERO NE PDGF BB A phase I/II, m u lticentre, randomized, controlled, open label trial compari ng the efficacy and safety of two dose regimens of BioChaperone PDGF BB to becaplermin gel for the treatment of diabetic foot u lcer.
- "Evaluation of Safety and Efficacy of Hydroxychloroquine Sulfate as an Adjunct to Diet and exercise to Improve Glycemic Control in Type 2 Diabetes Patients Uncontrolled on Sulfonylurea + etformin Combination" with tudy Code: Ipca/HCQS/PIV-14.
- 6. Study GOAL: Study of clinical and non clinical predictive factors for achieving glycemic control in people with type 2 diabetes in real clinical practice.
- 7. Effect and safety of semaglutide 2.4 mg once-weekly in subjects with overweight or obesity and type 2 diabetes.

- 8. ATOS I A Toujeo ® Observational Study
- A 12 month prospective observational study assessing the real world clinical effectiveness, safety and health economic benefits of Toujeo ® initiation after oral antidiabetic drug failure in insulin natve patients with type 2 diabetes mellitus
  - 9. Study Title: A Label extension, Randomized, Double Blind, Placebo Controlled, Multicentre, Single Dose, Phase III Study Assessing the Efficacy and Safety of Peri-ulcer Administration of stempeucel® (Adult Human Bone arrow Derived, Cultured, Pooled, Allogeneic Mesenchymal Stromal Cells) in Patients with Non-Healing Diabetic Foot Ulcer.
  - 10. The clinical trial "An observational, Cross sectional Study to assess the Prevalence of Heart Failure in Type 2 Diabetes Patients in India. Study Code: D1843R00300"
  - 11. The clinical trial "A Label extension, Randomized, Double Blind, Placebo Controlled, Multicentre, Single Dose, Phase III Study Assessing the Efficacy and Safety of Peri- ulcer Administration of stempeucel® (Adult Human Bone Marrow Derived, Cultured, Pooled, Allogeneic Mesenchymal Stromal Cells) in Patients with Non-Healin g Diabetic Foot Ulcer.
  - 12. The clinical trial "Ref: I8F- MC-GPHK: Efficacy and Safety of Tirzepatide Once Weekly in Participants without Type 2 Diabetes Who Have Obesity or are Overweight with Weight- Related Comorbidities: A Randomized, Double-Blind, Placebo- Controlled Trial(SURMOUNT 1)"

CAREER HIGHLIGHTS: Clinical Podiatrists since last 15 years.

Trained the paramedics on field of podiatry.

Retha Basak Strivastava 169

21



## **NIDA Clinical Trials Network**

### **Certificate of Completion**

is hereby granted to

### **GHANSHYAM GOYAL**

to certify your completion of the six-hour required course on:

### **GOOD CLINICAL PRACTICE**

| MODULE: | STATUS: |
|-------------------------------------|---------|
| Introduction | N/A |
| Institutional Review Boards | Passed |
| Informed Consent | Passed |
| Confidentiality & Privacy | Passed |
| Participant Safety & Adverse Events | Passed |
| Quality Assurance | Passed |
| The Research Protocol | Passed |
| Documentation & Record-Keeping | Passed |
| Research Misconduct | Passed |
| Roles & Responsibilities | Passed |
| Recruitment & Retention | Passed |
| Investigational New Drugs | Passed |

Course Completion Date: 13 May 2022 CTN Expiration Date: 13 May 2025

Eve Gelstrom

Eve Jelstrom, Principal Investigator NDAT CTN Clinical Coordinating Center

Good Clinical Practice, Version 5, effective 03-Mar-2017

This training has been funded in whole or in part with Federal funds from the National Institute on Drug Abuse, National Institutes of Health, Department of Health and Human Services, under Contract No. HHSN27201201000024C.



## NIDA Clinical Trials Network

## **Certificate of Completion**

is hereby granted to

## **REKHA BASAK SRIVASTAVA**

to certify your completion of the six-hour required course on:

### **GOOD CLINICAL PRACTICE**

| MODULE: | | STATUS: |
|-------------------------------------|---|---------|
| Introduction | | N/A |
| Institutional Review Boards | | Passed |
| Informed Consent | | Passed |
| Confidentiality & Privacy | * | Passed |
| Participant Safety & Adverse Events | | Passed |
| Quality Assurance | | Passed |
| Quality Assurance | | Passed |
| The Research Protocol | | Passed |
| Documentation & Record-Keeping | | Passed |
| Research Misconduct | | |
| Roles & Responsibilities | | Passed |
| Recruitment & Retention | | Passed |
| Investigational New Drugs | | Passed |

Course Completion Date: 23 December 2022 CTN Expiration Date: 23 December 2025

Eve Jelstrom

Eve Jelstrom, Principal Investigator NDAT CTN Clinical Coordinating Center

Good Clinical Practice, Version 5, effective 03-Mar-2017

This training has been funded in whole or in part with Federal funds from the National Institute on Drug Abuse, National Institutes of Health, Department of Health and Human Services, under Contract No. HH5N27201201000024C.



### WEST BENGAL MEDICAL COUNCIL

Constituated by the Govt. of West Bengal under Bengal Medical Act, 1914

IB - 196, Sector - III, Salt Lake, Kolkata – 700 106, West Bengal

### **Updated Registration Certificate - 2022**

Registration No.

: 47253 dated 16-06-1989

Name

: GOYAL

DR. GHAN SHYAM

Father's Name

SHAREWAN KUMAR GOYAL

Sex

: MALE

Address :

Permanent

IB - 127, SECTOR - III,

SALT LAKE CITY, PO: BIDHANNAGAR KOLKATA 700106 WEST BENGAL INDIA

Present

: IB - 127, SECTOR - III,

SALT LAKE CITY, PO: BIDHANNAGAR KOLKATA 700106 WEST BENGAL INDIA

Qualification: Basic

: M B B S (Rajasthan University), 1985

Additional

M D ( Genl. Med. ) ( Rajasthan University) , 1988

[Regd. on 11-01-2019]

202

Signature of Applicant Full:

lishm -

Specimen:

S. & hmm

Registrar, WBMC

**VALID TILL 31.12.2026** 

anas Karsale

